CLINICAL TRIAL: NCT05083910
Title: Randomized Controlled Comparison of Blood Loss in Patients Who Received Oxytocin Infusion, Oxytocin Infusion, and Intrauterine Misoprostol and Carbetocin During Cesarean Delivery
Brief Title: Randomization of Oxytocin, Oxytocin+Intrauterine Misoprostol and Carbetocin During C-section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20.5.2021-E.16677
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Postpartum Hemorrhage
Keywords: postpartum hemorrhage; oxytocin; misoprostol; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin Group (Experimental): The oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered immediately after clamping the umbilical cord
  Interventions: Drug: I.V Oxytocin administration
- Oxytocin+Intrauterine Misoprostol (Experimental): The oxytocin infusion was administered immediately after clamping the umbilical cord and misoprostol tablet (400 mg) was placed into uterine cavity at the fundus after delivery of the placenta and swabbing the cavity
  Interventions: Drug: I.V Oxytocin administration
- Carbetocin (Experimental): 100-mg carbetocin was intravenously administered immediately after birth of the baby
  Interventions: Drug: I.V Oxytocin administration

INTERVENTIONS:
Drug: I.V Oxytocin administration — Group I: Oxytocin( the oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered immediately after clamping the umbilical cord). Group II:oxytocin plus intrauterine misoprostol (the oxytocin infusion was administered immediately after clamping the umbilical cord and misoprostol tablet (400 mg) was placed into uterine cavity at the fundus after delivery of the placenta and swabbing the cavity. Group III:100-mg carbetocin was intravenously administered immediately after birth of the baby.
  Other Names: I.v Oxytocin+intrauterine misoprostol; I.V carbetocin administration

SUMMARY:
Postpartum haemorrhage (PPH) remains an important cause of maternal morbidity and mortality and it accounts for approximately 25% of all deaths worldwide. Drugs such as oxytocin, carbetocin, misoprostol, prostaglandin F2a and methylergonovine have been tested for bleeding control during and after cesarean section. Oxytocin is the most widely used agent for the prevention of postpartum hemorrhage.The primary aim of this study is to reduce the mean blood loss during cesarean section.In this study, the investigators planned to compare peroperative and postoperative blood loss levels by giving oxytocin alone to the 1st group, oxytocin and intrauterine misoprostol to the 2nd group, and carbetocin to the 3rd group of patients who were randomly divided into 3 groups.In this study, we aimed to compare the efficacy of oxytocin, misoprostol and carbetocin in preventing uterine blood loss during cesarean section.

DETAILED DESCRIPTION:
Our prospective, randomized controlled study was conducted at the Department of Obstetrics and Gynecology of Bezmialem University Hospital between July and November 2021. The study protocol was approved by the Ethical Committee of the Medical Faculty of Bezmialem University. Written informed consent was obtained from all patients. We included a total of 156 women between 18 and 40 years of age who underwent a primary cesarean section or old 1 cesarean section under spinal anesthesia at term single pregnancy with an American Society of Anesthesiology physical status of I or II. This trial was designed and reported according to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

The patients included in this study were randomly divided into three groups by random allocation using a computer-generated random number. Group I: Oxytocin(Synpitan forte®; Deva Pharma, Istanbul, Turkey) (n = 52 )( the oxytocin infusion consisting of 20 IU dissolved in 500 mL of normal 0.9 % sodium chloride solution and infused at a rate of 125 mL/h was administered immediately after clamping the umbilical cord). Group II: (n =52) oxytocin plus intrauterine misoprostol (Synpitan forte®; Deva Pharma, Istanbul, Turkey) (the oxytocin infusion was administered immediately after clamping the umbilical cord and misoprostol tablet (400 mg) was placed into uterine cavity at the fundus after delivery of the placenta and swabbing the cavity. Group III: (n =52) 100-mg carbetocin (Synpitan forte®; Deva Pharma, Istanbul, Turkey) was intravenously administered immediately after birth of the baby. All surgeries were performed by the same team of two surgeons.. The collected data were age, prepregnancy body mass index (BMI), gravida, parity, indication of cesarean section, gestational age at birth, Apgar scores at 1 and 5 min, birth weight, neonatal intensive care unit (NICU) admission, the preoperative hemoglobin and hematocrit concentrations, the change in the hemoglobin and hematocrit concentrations (difference between preoperative and postoperative levels), operating time, intraoperative blood loss.

In this study, the investigators aimed to compare the efficacy of oxytocin, misoprostol and carbetocin in preventing uterine blood loss during cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy greater than 37 weeks
* Pregnant women between the ages of 18-40 Volunteer

Exclusion Criteria:

* Clinical diagnosis of Gestational diabetes
* Clinical diagnosis of Gestational hypertension
* Clinical diagnosis of preeclampsia
* Clinical diagnosis of Placenta previa,
* Clinical diagnosis of abruptio placenta
* Conditions that cause excessive distention of the uterus (multiple pregnancies, severe polyhydramnios, fetal macrosomia, large fibroids displacing the cavity) Thrombophilia disorders, anticoagulation therapy History of major abdominal surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 156 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-22 (Actual)

PRIMARY OUTCOMES:
Hemogram status | Postoperative 8th hour
  Postoperative hemogram status

SECONDARY OUTCOMES:
Blood Transfusion | Postoperative 24th hour
  Number of patients needing Blood Transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Kıran, MD, Study Chair — Bezmialem Vakif University
Locations (2):
- Turkey (Türkiye) (2):
  - Bezmialem Vakif University, Istanbul, Istanbulk
  - Bezmialem Vakif University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibrahim ZM, Sayed Ahmed WA, Abd El-Hamid EM, Taha OT, Elbahie AM. Carbetocin versus oxytocin for prevention of postpartum hemorrhage in hypertensive women undergoing elective cesarean section. Hypertens Pregnancy. 2020 Aug;39(3):319-325. doi: 10.1080/10641955.2020.1768268. Epub 2020 May 18. PMID 32421401
- [Result] Takmaz T, Ozcan P, Sevket O, Karasu AFG, Islek SH, Halici BNA. Less Blood Loss by Earlier Oxytocin Infusion in Cesarean Sections? A Randomized Controlled Trial. Z Geburtshilfe Neonatol. 2020 Oct;224(5):275-280. doi: 10.1055/a-1108-2017. Epub 2020 Mar 2. PMID 32120445
- [Result] Bahadur A, Khoiwal K, Bhattacharya N, Chaturvedi J, Kumari R. The effect of intrauterine misoprostol on blood loss during caesarean section. J Obstet Gynaecol. 2019 Aug;39(6):753-756. doi: 10.1080/01443615.2019.1581743. Epub 2019 Apr 22. PMID 31010345